CLINICAL TRIAL: NCT00793377
Title: A Randomized, Multicenter, Open Phase III Study Comparing a Dose-Intensified 8 Week Schedule of Adriamycin and Docetaxel (ADOC) With a Sequential 24 Week Schedule of Adriamycin/Cyclophosphamide Followed by Docetaxel (AC-DOC) Regimen as Preoperative Therapy in Patients With Operable Carcinoma of the Breast (T2-3 N0-2 M0)
Brief Title: Neoadjuvant Doxorubicin/Cyclophosphamide Followed by Docetaxel (AC-Doc) Versus Dose-Dense Doxorubicin and Docetaxel (ADoc) in Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GBG Forschungs GmbH (Other)
Collaborators: German Adjuvant Breast Cancer Group (Other)
Responsible Party: Prof. Dr. G. v. Minckwitz, GBG Forschungs GmbH
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: Gepar-Duo
Record Dates: First submitted 2008-11-17; First posted 2008-11-19 (Estimated); Last update posted 2008-11-19 (Estimated); Status verified 2008-11

CONDITIONS: Primary Breast Cancer
MeSH Terms: interventions — Doxorubicin; Docetaxel; Tamoxifen; Cyclophosphamide

ARMS (2):
- ADOC x 4 + Tam 20 (Experimental): Adriamycin will be given at a dose of 50 mg/m2 and docetaxel at a dose of 75 mg/m2 every 14 days for four cycles. Adriamycin will be administered as a short i.v. infusion over 15 minutes, followed immediately by a 1-hour infusion of docetaxel diluted in 250 mL NaCl. Tamoxifen 20 mg is given once daily for five years to all patients, starting with the first day of chemotherapy.
  Interventions: Drug: Adriamycin (Doxorubicin), Docetaxel, Tamoxifen
- AC x 4 - Doc x 4 + Tam 20 (Experimental): Adriamycin will be given at a dose of 60 mg/m2 and cyclophosphamide at a dose of 600 mg/m2 every 21 days for four cycles. Thereafter, docetaxel at a dose of 100 mg/m2 is given every 21 days for four cycles. Tamoxifen 20 mg is given once daily for five years to all patients, starting with the first day of chemotherapy
  Interventions: Drug: Adriamycin (Doxorubicin), Docetaxel, Tamoxifen, Cyclophosphamid

INTERVENTIONS:
Drug: Adriamycin (Doxorubicin), Docetaxel, Tamoxifen — Adriamycin will be given at a dose 50 mg/m2 and docetaxel at a dose of 75 mg/m2 every 14 days for four cycles.Tamoxifen 20 mg is given once daily for five years to all patients, starting with the first day of chemotherapy.
  Arms: ADOC x 4 + Tam 20
Drug: Adriamycin (Doxorubicin), Docetaxel, Tamoxifen, Cyclophosphamid — Adriamycin will be given at a dose of 60 mg/m2 and cyclophosphamide at a dose of 600 mg/m2 every 21 days for four cycles. Thereafter, docetaxel at a dose of 100 mg/m2 is given every 21 days for four cycles. Tamoxifen 20 mg is given once daily for five years to all patients, starting with the first day of chemotherapy.
  Arms: AC x 4 - Doc x 4 + Tam 20

SUMMARY:
The primary objective of this trial is to compare the rate of pathologically complete remissions achieved using a preoperative dose-intensified 8 week therapy consisting of adriamycin and docetaxel with a preoperative sequential 24 week regimen consisting of adriamycin/cyclophosphamide followed by docetaxel, in patients with operable carcinoma of the breast. Secondary aims are to assess disease-free and overall survival, the rate of complete and partial responses by palpation and imaging methods, the rate of breast-conserving operations, and the toxicity of the two chemotherapy regimens.

Women meeting the following criteria will be eligible for the study: those with operable breast cancer (T2-3 N0-2 M0), with the diagnosis histologically confirmed by biopsy, and measurable disease on mammography or sonography or breast MRI (the most appropriate method should be chosen by the investigator). After the patients have given written informed consent, they will be randomly assigned to the study treatments. Patients in group I will receive four cycles of combination chemotherapy consisting of adriamycin 50 mg/m2 (15 min i.v. infusion) and docetaxel 75 mg/m2 (1 h i.v. infusion) repeated every 14 days, followed by surgery 9-10 weeks after the start of therapy. Patients in group II will receive four cycles of adriamycin 60 mg/m2 (15 min i.v.) and cyclophosphamide 600 mg/m2 (1 h i.v.) every three weeks, followed by four cycles of docetaxel 100 mg/m2 (1 h i.v.) every three weeks. Surgery will be performed during week 25 or 26. Patients in both groups will additionally receive oral doses of tamoxifen 20 mg once daily for 5 years, starting on the first day of chemotherapy. Surgery will consist of removal of the remaining tumor (breast-conserving resection or mastectomy) and axillary dissection (Sentinel node biopsy is allowed if the patient is involved in a randomized trial. Radiotherapy is applicated according to standard proceedings of participating center. A second randomization for additional versus no additional postoperative chemotherapy is recommended in ypN+ disease. Patients with disease progression during preoperative therapy, chemotherapy can be stopped and surgery can be performed immediately.

ELIGIBILITY:
Inclusion Criteria:

* Pre-study screening performed according to section 7.1
* Unilateral primary carcinoma of the breast, confirmed histologically by core or tru-cut biopsy. Fine-needle aspiration is not sufficient. Incisional biopsy is only allowed if less than 20% of the tumor is excised.
* Two-dimensionally measurable (mammography, ultrasound, or MRI) breast tumor
* Primary tumor >= 2 cm in largest diameter by either palpation, sonography or mammography, or breast MRI. In patients with multifocal or multicentric breast cancer, the largest lesion should be measured.
* No evidence of distant metastases
* Life expectancy of at least 10 years, disregarding the diagnosis of cancer.
* Karnofsky index >= 70%.
* Age 18 years or older.
* Adequate hematological, renal, and hepatic function (WBC > 4000, platelets > 100 000, bilirubin, serum creatinine and transaminases within 1.5 × upper normal range).
* Evidence of normal cardiac function (with or without medication) from the patient history and from electrocardiography. Normal function is confirmed by echocardiography or multiple gated acquisition (MUGA) scan.
* Negative pregnancy test and appropriate nonhormonal contraception in fertile women. Intrauterine pessaries with progestogens are allowed.
* Written informed consent and assumed compliance for therapy and follow up of the patients.
* Consent of patient, pathologist and investigator to supply tumor material of biopsy and surgery for central pathologic evaluation and examination of predictive factors.

Exclusion Criteria:

* Locally advanced (stage T4), bilateral, metastatic, or inflammatory breast cancer. If one of these conditions is suspected, it has to be excluded before enrollment into study.
* Previous treatment for breast cancer, including surgery, radiation, cytotoxic, or endocrine treatments.
* Previous malignancy other than breast cancer or noninvasive breast cancer if the disease-free interval is less than 10 years.
* Previous cytotoxic treatment for any condition.
* Preexisting neurotoxicity greater than grade II.
* Active infection or other significant illness that could influence the tolerability of treatment.
* Current treatment with sex hormones (treatment has to be discontinued before the start of systemic therapy).
* Psychiatric illness or drug addiction that would preclude obtaining informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 913 (Actual)
Dates: Study Completion 2001-09 (Actual)

PRIMARY OUTCOMES:
Pathological locoregional complete tumor response (pCR) between both arms | 3 years

SECONDARY OUTCOMES:
Survival Local tumor response by palpation (cRR=cCR+cPR) Local tumor response by best imaging method (iRR=iCR+iPR) Response of axillary lymphnodes (NR) Breast conservation therapy (BCT) Toxicity | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- German Breast Group, Neu-Isenburg, Hesse, Germany

REFERENCES:
- [Background] Jackisch C, von Minckwitz G, Eidtmann H, Costa SD, Raab G, Blohmer JU, Schutte M, Gerber B, Merkle E, Gademann G, Lampe D, Hilfrich J, Tulusan AH, Caputo A, Kaufmann M. Dose-dense biweekly doxorubicin/docetaxel versus sequential neoadjuvant chemotherapy with doxorubicin/cyclophosphamide/docetaxel in operable breast cancer: second interim analysis. Clin Breast Cancer. 2002 Oct;3(4):276-80. doi: 10.3816/cbc.2002.n.031. PMID 12425756
- [Result] Loibl S, von Minckwitz G, Raab G, Blohmer JU, Dan Costa S, Gerber B, Eidtmann H, Petrich S, Hilfrich J, Jackisch C, du Bois A, Kaufmann M. Surgical procedures after neoadjuvant chemotherapy in operable breast cancer: results of the GEPARDUO trial. Ann Surg Oncol. 2006 Nov;13(11):1434-42. doi: 10.1245/s10434-006-9011-2. Epub 2006 Sep 17. PMID 16983592
- [Result] von Minckwitz G, Raab G, Caputo A, Schutte M, Hilfrich J, Blohmer JU, Gerber B, Costa SD, Merkle E, Eidtmann H, Lampe D, Jackisch C, du Bois A, Kaufmann M. Doxorubicin with cyclophosphamide followed by docetaxel every 21 days compared with doxorubicin and docetaxel every 14 days as preoperative treatment in operable breast cancer: the GEPARDUO study of the German Breast Group. J Clin Oncol. 2005 Apr 20;23(12):2676-85. doi: 10.1200/JCO.2005.05.078. PMID 15837982
- [Derived] von Minckwitz G, Untch M, Blohmer JU, Costa SD, Eidtmann H, Fasching PA, Gerber B, Eiermann W, Hilfrich J, Huober J, Jackisch C, Kaufmann M, Konecny GE, Denkert C, Nekljudova V, Mehta K, Loibl S. Definition and impact of pathologic complete response on prognosis after neoadjuvant chemotherapy in various intrinsic breast cancer subtypes. J Clin Oncol. 2012 May 20;30(15):1796-804. doi: 10.1200/JCO.2011.38.8595. Epub 2012 Apr 16. PMID 22508812
- [Derived] Darb-Esfahani S, Loibl S, Muller BM, Roller M, Denkert C, Komor M, Schluns K, Blohmer JU, Budczies J, Gerber B, Noske A, du Bois A, Weichert W, Jackisch C, Dietel M, Richter K, Kaufmann M, von Minckwitz G. Identification of biology-based breast cancer types with distinct predictive and prognostic features: role of steroid hormone and HER2 receptor expression in patients treated with neoadjuvant anthracycline/taxane-based chemotherapy. Breast Cancer Res. 2009;11(5):R69. doi: 10.1186/bcr2363. PMID 19758440
- See also: Related Info — http://germanbreastgroup.de